CLINICAL TRIAL: NCT00162097
Title: Pharmacokinetics of Efavirenz During Treatment of HIV-1 Infected Subjects With Hepatic Impairment.
Brief Title: Pharmacokinetics of Efavirenz in HIV-1 Infected Subjects With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI266-917
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Results first posted 2010-08-25 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: HIV Infections; Hepatic Impairment
MeSH Terms: conditions — HIV Infections | interventions — efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- EFV600mg Participants With Mild Hepatic Impairment (Experimental)
  Interventions: Drug: efavirenz containing antiretroviral regimen
- EFV600mg Participants With Moderate Hepatic Impairment (Experimental)
  Interventions: Drug: efavirenz containing antiretroviral regimen
- EFV600mg Participants With Severe Hepatic Impairment (Experimental)
  Interventions: Drug: efavirenz containing antiretroviral regimen
- EFV600mg Participants With Normal Hepatic Function (Active Comparator)
  Interventions: Drug: efavirenz containing antiretroviral regimen

INTERVENTIONS:
Drug: efavirenz containing antiretroviral regimen — Capsule or Tablet, Oral, once daily for 2 days
  Other Names: Sustiva; BMS-561525
  Arms: EFV600mg Participants With Mild Hepatic Impairment
Drug: efavirenz containing antiretroviral regimen — Capsule or Tablet, Oral, once daily for 2 days
  Other Names: Sustiva; BMS-561525
  Arms: EFV600mg Participants With Moderate Hepatic Impairment
Drug: efavirenz containing antiretroviral regimen — Capsule or Tablet, Oral, once daily for 2 days
  Other Names: Sustiva; BMS-561525
  Arms: EFV600mg Participants With Severe Hepatic Impairment
Drug: efavirenz containing antiretroviral regimen — Capsule or Tablet, Oral, once daily for 2 days
  Other Names: Sustiva; BMS-561525
  Arms: EFV600mg Participants With Normal Hepatic Function

SUMMARY:
The purpose of the study was to assess the steady-state pharmacokinetics (PK) of efavirenz (EFV) in human immunodeficiency virus type 1 (HIV-1) infected subjects on stable antiretroviral regimens containing EFV, and having selected degrees of hepatic impairment or normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection with or without Hepatitis B or C infection
* Stable antiretroviral regimen containing efavirenz and nucleoside/nucleotide reverse transcriptase inhibitors (NRTI) for at least 1 month
* Mild, moderate or severe hepatic impairment with hepatic cirrhosis

Exclusion Criteria:

* Acute flare of hepatitis
* Positive pregnancy test for a female
* Significant acute medical illness in past 2 months
* Use of agents known to significantly affect liver metabolism
* Change in medications to treat a chronic disease in the past 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2004-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (3):
  - Johns Hopkins University School Of Medicine, Baltimore, Maryland
  - Uthscsa, San Antonio, Texas
  - Virginia Commonwealth University Health Systems, Richmond, Virginia
- Local Institution, Milan, Italy

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 21 participants were enrolled in the study; 5 discontinued prior to study drug administration (1 adverse event, 1 enrollment completed, 1 screen failure, 1 no longer met study criteria and 1 withdrew consent).
Groups:
- EFV600mg Participants With Mild Hepatic Impairment: Participants were administered a dose of 600 mg once daily (capsules or tablets) of efavirenz, either in the morning (at approximately 9:00 AM) or before bed time (at approximately 9:00 PM), on an empty stomach. The duration of efavirenz administration was 2 days and participants were admitted to the clinical facility for this period. Mild hepatic impairment (grade A) is defined as a Child-Pugh (CP) total score of 5-6. The CP classification assesses 5 hepatic parameters (total serum bilirubin, serum albumin, prothrombin time, ascites and encephalopathy) on a scale of 1 (mild or none) to 3 (most severe). Total score range is 5 (mild) to 15 (severe).
- EFV600mg Participants With Moderate Hepatic Impairment: Participants were administered a dose of 600 mg once daily (capsules or tablets) of efavirenz, either in the morning (at approximately 9:00 AM) or before bed time (at approximately 9:00 PM), on an empty stomach. The duration of efavirenz administration was 2 days and participants were admitted to the clinical facility for this period. Moderate hepatic impairment (grade B) is defined as a CP total score of 7-9.
- EFV600mg Participants With Severe Hepatic Impairment: Participants were administered a dose of 600 mg once daily (capsules or tablets) of efavirenz, either in the morning (at approximately 9:00 AM) or before bed time (at approximately 9:00 PM), on an empty stomach. The duration of efavirenz administration was 2 days and participants were admitted to the clinical facility for this period. Participants who were on an off-label reduced dose of efavirenz (eg, 400 mg) continued on the reduced dose. Severe hepatic impairment (grade C) is defined as a CP total score of 10-15.
- EFV600mg Participants With Normal Hepatic Function: Participants were administered a dose of 600 mg once daily (capsules or tablets) of efavirenz either in the morning (at approximately 9:00 AM) or before bed time (at approximately 9:00 PM) on an empty stomach. The duration of efavirenz administration was 2 days when participants were admitted to the clinical facility. Participants were enrolled after at least 6 participants with hepatic impairment had completed. One participant enrolled twice in the study and is hence counted twice in this group
Period: Overall Study
Arm/Group | EFV600mg Participants With Mild Hepatic Impairment | EFV600mg Participants With Moderate Hepatic Impairment | EFV600mg Participants With Severe Hepatic Impairment | EFV600mg Participants With Normal Hepatic Function
Started | 6 (Treated on Day 1) | 2 (Treated on Day 1) | 1 (Treated on Day 1) | 7 (Treated on Day 1. One participant enrolled twice in the study and is hence counted twice)
Completed | 6 | 2 | 1 | 6
Not Completed | 0 | 0 | 0 | 1
Not completed — Participant no longer met study criteria | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EFV600mg Participants With Mild Hepatic Impairment | EFV600mg Participants With Moderate Hepatic Impairment | EFV600mg Participants With Severe Hepatic Impairment | EFV600mg Participants With Normal Hepatic Function | Total
Number analyzed (Participants) | 6 | 2 | 1 | 7 | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 50 (11) | 51 (1) | 47 | 49 (4) | 49 (7)
Age, Customized [Number; unit: participants]
  < 65 years | 5 | 2 | 1 | 7 | 15
  >= 65 years | 1 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 1 | 0 | 5
  Male | 2 | 2 | 0 | 7 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 5 | 2 | 0 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian | 1 | 0 | 0 | 0 | 1
  Black | 3 | 1 | 0 | 5 | 9
  White | 2 | 1 | 0 | 2 | 5
  Hispanic/Latino | 0 | 0 | 1 | 0 | 1
Body mass index (BMI) Continuous [Mean (Standard Deviation); unit: kg/m^2] — BMI is defined as the individual's body weight divided by the square of his or her height.
  kg/m^2 | 26.3 (3.7) | 24.6 (0.1) | 24.0 | 22.8 (2.2) | 24.4 (3.0)
Height Continuous [Mean (Standard Deviation); unit: cm] | 165.5 (11.9) | 173.4 (3.7) | 160.0 | 175.6 (7.2) | 170.6 (10.0)
Weight, Continuous [Mean (Standard Deviation); unit: kilogram] | 71.5 (7.2) | 73.9 (2.9) | 61.5 | 70.4 (9.6) | 70.7 (7.9)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: Cmax was obtained directly from the concentration-time data.
Time Frame: Blood samples were collected at time 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose, relative to administration of PM or AM dose.
Population: The analysis was performed per protocol.
Measure: Geometric Mean (Full Range); unit: micrograms (mcg)/mL
Arm/Group | EFV600mg Participants With Mild Hepatic Impairment | EFV600mg Participants With Moderate Hepatic Impairment | EFV600mg Participants With Severe Hepatic Impairment | EFV600mg Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 2 | 1 | 6
micrograms (mcg)/mL | 5.303 [2.730 to 16.000] | 8.964 [4.900 to 16.400] | 6.750 [6.750 to 6.750] | 6.515 [2.680 to 25.300]

2. Secondary Outcome: Number of Participants Who Died or Experienced Other Serious Adverse Events (SAEs)
Description: An SAE was defined as any adverse event (AE) occurring at any dose that; resulted in death; was life threatening; resulted in a persistent or significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; was a cancer; or was an overdose.
Time Frame: From screening (within 21 days of Day 1 dosing) to the study discharge day (Day 2 for AM dosing or Day 3 for PM dosing). Participants were monitored for SAEs up to 30 days after study discharge.
Population: All data from participants who signed the informed consent and enrolled in the study is included in the data set used for evaluating SAEs.
Measure: Number; unit: Participants
Groups:
- Participants With Mild Hepatic Impairment: Participants were administered a dose of 600 mg once daily (capsules or tablets) of efavirenz, either in the morning (at approximately 9:00 AM) or before bed time (at approximately 9:00 PM), on an empty stomach. The duration of efavirenz administration was 2 days and participants were admitted to the clinical facility for this period. Mild hepatic impairment (grade A) is defined as a Child-Pugh (CP) total score of 5-6. The CP classification assesses 5 hepatic parameters (total serum bilirubin, serum albumin, prothrombin time, ascites and encephalopathy) on a scale of 1 (mild or none) to 3 (most severe). Total score range is 5 (mild) to 15 (severe).
- Participants With Moderate Hepatic Impairment: Participants were administered a dose of 600 mg once daily (capsules or tablets) of efavirenz, either in the morning (at approximately 9:00 AM) or before bed time (at approximately 9:00 PM), on an empty stomach. The duration of efavirenz administration was 2 days and participants were admitted to the clinical facility for this period. Moderate hepatic impairment (grade B) is defined as a CP total score of 7-9.
- Participants With Severe Hepatic Impairment: Participants were administered a dose of 600 mg once daily (capsules or tablets) of efavirenz, either in the morning (at approximately 9:00 AM) or before bed time (at approximately 9:00 PM), on an empty stomach. The duration of efavirenz administration was 2 days and participants were admitted to the clinical facility for this period. Participants who were on an off-label reduced dose of efavirenz (eg, 400 mg) continued on the reduced dose. Severe hepatic impairment (grade C) is defined as a CP total score of 10-15.
- Participants With Normal Hepatic Function: Participants were administered a dose of 600 mg once daily (capsules or tablets) of efavirenz either in the morning (at approximately 9:00 AM) or before bed time (at approximately 9:00 PM) on an empty stomach. The duration of efavirenz administration was 2 days when participants were admitted to the clinical facility. Participants were enrolled after at least 6 participants with hepatic impairment had completed. One participant enrolled twice in the study and is hence counted twice in this group
- Participants Not Dosed: Participants were enrolled in the study and discontinued prior to study drug administration
Arm/Group | Participants With Mild Hepatic Impairment | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment | Participants With Normal Hepatic Function | Participants Not Dosed
Number analyzed (Participants) | 6 | 2 | 1 | 7 | 5
Participants
  Deaths | 0 | 0 | 0 | 0 | 1
  Other Serious Adverse Events | 0 | 0 | 0 | 0 | 1

3. Primary Outcome: Minimum Plasma Concentration (Cmin)
Description: Cmin was obtained directly from the concentration-time data.
Time Frame: as for outcome 1
Population: The analysis was performed per protocol.
Measure: Geometric Mean (Full Range); unit: mcg/mL
Arm/Group | EFV600mg Participants With Mild Hepatic Impairment | EFV600mg Participants With Moderate Hepatic Impairment | EFV600mg Participants With Severe Hepatic Impairment | EFV600mg Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 2 | 1 | 6
mcg/mL | 2.599 [0.688 to 11.500] | 4.885 [1.850 to 12.900] | 3.780 [3.780 to 3.780] | 2.405 [0.611 to 17.900]

4. Primary Outcome: Area Under the Plasma Concentration-time Curve Over the Dosing Interval of 24 Hours (AUC[TAU])
Description: The AUC(TAU), from time 0 to the time of the last measurable concentration (t), was calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Population: The analysis was performed per protocol.
Measure: Geometric Mean (Full Range); unit: mcg*h/mL
Arm/Group | EFV600mg Participants With Mild Hepatic Impairment | EFV600mg Participants With Moderate Hepatic Impairment | EFV600mg Participants With Severe Hepatic Impairment | EFV600mg Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 1 | 1 | 6
mcg*h/mL | 83.422 [29.84 to 323.06] | 75.425 [75.425 to 75.425] | 101.912 [101.912 to 101.912] | 93.516 [36.51 to 486.43]

5. Secondary Outcome: Number of Participants Who Experienced AEs
Description: AEs were defined as any new untoward medical occurrences or worsening of a pre-existing medical condition in a participant administered a medicinal product, whether or not considered related to the medicinal product.
Time Frame: From screening (within 21 days of Day 1 dosing) to the study discharge day (Day 2 for AM dosing or Day 3 for PM dosing).
Population: All participants who received study drug on Day 1 were included in the analysis.
Measure: Number; unit: participants
Arm/Group | EFV600mg Participants With Mild Hepatic Impairment | EFV600mg Participants With Moderate Hepatic Impairment | EFV600mg Participants With Severe Hepatic Impairment | EFV600mg Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 2 | 1 | 7
participants | 1 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants Who Experienced AEs Leading to Study Drug Discontinuation
Description: AEs were defined as any new untoward medical occurrences or worsening of a pre-existing medical condition in a participant administered a medicinal product, whether or not considered related to the medicinal product. Participants who discontinued the study due to an AE were recorded.
Time Frame: From screening (within 21 days of Day 1 dosing) to the study discharge day (Day 2 for AM dosing or Day 3 for PM dosing).
Population: All participants who received study drug on Day 1 were included in the analysis.
Measure: Number; unit: participants
Arm/Group | EFV600mg Participants With Mild Hepatic Impairment | EFV600mg Participants With Moderate Hepatic Impairment | EFV600mg Participants With Severe Hepatic Impairment | EFV600mg Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 2 | 1 | 7
participants | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Marked Abnormalities (MAs) in Hematology Measurements
Description: MAs are laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. The following hematology MA definitions specify the criteria for the data presented. Low platelet count: <0.85 x lower limit of normal (LLN) (or if pre-treatment value <LLN, then <0.85 x pre-treatment value). Low leukocytes: <0.9 x LLN (or if pre-treatment value <LLN, then <0.85 x pre-treatment value. If pre-treatment value >upper limit of normal [ULN], then <LLN). Low neutrophils+bands (absolute): <=1.500 10^3 cells/microliter (uL). Low lymphocytes (absolute): <0.750 10^3 cells/uL.
Time Frame: Throughout study, from screening (within 21 days of Day 1 dosing) through Day 3.
Population: All participants who received study drug on Day 1 and were evaluated for these measures.
Measure: Number; unit: participants
Arm/Group | EFV600mg Participants With Mild Hepatic Impairment | EFV600mg Participants With Moderate Hepatic Impairment | EFV600mg Participants With Severe Hepatic Impairment | EFV600mg Participants With Normal Hepatic Function
Number analyzed (Participants) | 5 | 2 | 1 | 7
participants
  Low platelet count | 0 | 1 | 0 | 0
  Low leukocytes | 1 | 0 | 0 | 1
  Low neutrophils+bands (absolute) | 1 | 2 | 1 | 0
  Low lymphocytes (absolute) | 0 | 0 | 1 | 0

8. Secondary Outcome: Number of Participants With Serum Chemistry MAs
Description: MAs are laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. The following serum chemistry MA definitions specify the criteria for MAs in the data presented. High bilirubin (total): >1.1 x ULN (or if pre-treatment value >ULN, then >1.25 x pre-treatment value). High creatinine: >1.33 x pre-treatment value. Low albumin: <0.9 x LLN (or if pre-treatment value <LLN, then <0.9 x pre-treatment value). High amylase (total): >2 x pre-treatment value.
Time Frame: Throughout study, from screening (within 21 days of Day 1 dosing) through Day 3.
Population: All participants who received study drug on Day 1 were included in the analysis. The 'n' signifies those participants who received study drug and were evaluated for this measure, for each group respectively.
Measure: Number; unit: participants
Arm/Group | EFV600mg Participants With Mild Hepatic Impairment | EFV600mg Participants With Moderate Hepatic Impairment | EFV600mg Participants With Severe Hepatic Impairment | EFV600mg Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 2 | 1 | 7
participants
  High bilirubin (total) (n = 5, 1, 1, 7) | 1 | 0 | 0 | 0
  High creatinine (n = 5, 1, 1, 7) | 0 | 0 | 0 | 1
  Low albumin (n = 5, 1, 1, 7) | 0 | 1 | 0 | 0
  High amylase (total) (n = 5, 1, 0, 7) | 0 | 0 | 0 | 1

9. Secondary Outcome: Number of Participants With Urinalysis MAs
Description: MAs are laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. The following urinalysis MA definitions specify the criteria for MAs in the data presented. The presence of white blood cells (WBCs) and red blood cells (RBCs) in the urine was graded on a scale: 0 = no cells present (negative); trace =a small number of cells present; then 1+, 2+, 3+ and 4+, denoting increasingly "positive" urine results (ie, WBCs/RBCs present in the urine). The MA for both WBCs and RBCs was >= 2+ (or, if pre-treatment value >=2+, then >= 4+).
Time Frame: Throughout study, from screening (within 21 days of Day 1 dosing) through Day 3.
Population: All participants who received study drug on Day 1 and were evaluated for these measures.
Measure: Number; unit: participants
Arm/Group | EFV600mg Participants With Mild Hepatic Impairment | EFV600mg Participants With Moderate Hepatic Impairment | EFV600mg Participants With Severe Hepatic Impairment | EFV600mg Participants With Normal Hepatic Function
Number analyzed (Participants) | 5 | 1 | 1 | 7
participants
  White blood cells (WBCs) | 1 | 0 | 0 | 0
  Red blood cells (RBCs) | 1 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Identified Electrocardiogram (ECG) Abnormalities
Description: ECG abnormalities are findings that are clinically meaningful by the judgment of the investigator. A 12-lead ECG was performed and all ECG recordings were evaluated by the investigator. Abnormalities, if present at any study time point, were listed.
Time Frame: From screening (within 21 days of Day 1 dosing) to the study discharge day (Day 2 for AM dosing or Day 3 for PM dosing)
Population: All participants who received study drug on Day 1 were included in the analysis.
Measure: Number; unit: participants
Arm/Group | EFV600mg Participants With Mild Hepatic Impairment | EFV600mg Participants With Moderate Hepatic Impairment | EFV600mg Participants With Severe Hepatic Impairment | EFV600mg Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 2 | 1 | 7
participants | 3 | 1 | 0 | 5

11. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Description: Tmax was obtained directly from the concentration-time data.
Time Frame: as for outcome 1
Population: The analysis was performed per protocol.
Measure: Median (Full Range); unit: hours
Arm/Group | EFV600mg Participants With Mild Hepatic Impairment | EFV600mg Participants With Moderate Hepatic Impairment | EFV600mg Participants With Severe Hepatic Impairment | EFV600mg Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 2 | 1 | 6
hours | 1.765 [0.98 to 6.03] | 4.500 [3.00 to 6.00] | 1.000 [1.00 to 1.00] | 3.500 [2.00 to 6.00]

12. Secondary Outcome: Number of Participants With Clinically Meaningful Vital Signs Measures
Description: Vital signs were recorded throughout the study and included investigations related to body temperature, respiratory rate, seated blood pressure (systolic and diastolic), and heart rate. The investigator used his/her clinical judgement to decide whether or not abnormalities in vital signs were clinically meaningful.
Time Frame: From screening (within 21 days of Day 1 dosing) to the study discharge day (Day 2 for AM dosing or Day 3 for PM dosing)
Population: All participants who received study drug on Day 1 were included in the analysis.
Measure: Number; unit: participants
Arm/Group | EFV600mg Participants With Mild Hepatic Impairment | EFV600mg Participants With Moderate Hepatic Impairment | EFV600mg Participants With Severe Hepatic Impairment | EFV600mg Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 2 | 1 | 7
participants | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Abnormal Physical Examination Findings at Baseline (Screening and/or Day 1)
Description: The physical examination included an evaluation of the participant's height and body mass index (BMI) (at screening only), and weight. Abnormal physical examination are findings that are clinically meaningful by the judgment of the investigator
Time Frame: From screening (within 21 days of Day 1 dosing) to the study discharge day (Day 2 for AM dosing or Day 3 for PM dosing)
Population: All participants who received study drug on Day 1 were included in the analysis. Physical examination findings were not analysed at discharge.
Measure: Number; unit: participants
Arm/Group | EFV600mg Participants With Mild Hepatic Impairment | EFV600mg Participants With Moderate Hepatic Impairment | EFV600mg Participants With Severe Hepatic Impairment | EFV600mg Participants With Normal Hepatic Function
Number analyzed (Participants) | 6 | 2 | 1 | 7
participants | 5 | 2 | 1 | 5

ADVERSE EVENTS:
Description: One participant enrolled twice in the study in EFV600mg participants with normal hepatic function group and is hence counted twice in this group.
Arm/Group | EFV600mg Participants With Mild Hepatic Impairment | EFV600mg Participants With Moderate Hepatic Impairment | EFV600mg Participants With Severe Hepatic Impairment | EFV600mg Participants With Normal Hepatic Function | Not Dosed
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2 | 0/1 | 0/7 | 1/5
Other Adverse Events (participants affected / at risk) | 1/6 | 0/2 | 0/1 | 0/7 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EFV600mg Participants With Mild Hepatic Impairment (N=6) | EFV600mg Participants With Moderate Hepatic Impairment (N=2) | EFV600mg Participants With Severe Hepatic Impairment (N=1) | EFV600mg Participants With Normal Hepatic Function (N=7) | Not Dosed (N=5)
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
AIDS RELATED COMPLICATION (Infections and infestations) | 0 | 0 | 0 | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EFV600mg Participants With Mild Hepatic Impairment (N=6) | EFV600mg Participants With Moderate Hepatic Impairment (N=2) | EFV600mg Participants With Severe Hepatic Impairment (N=1) | EFV600mg Participants With Normal Hepatic Function (N=7) | Not Dosed (N=5)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early leading to a small number of participants treated and analyzed. Due to the small sample size, no conclusion could be made for participants with Child-Pugh scores B and C (moderate and severe hepatic impairment).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.